CLINICAL TRIAL: NCT01702077
Title: Neurofeedback of Activity in the Supplementary Motor Area for Tourette Syndrome
Brief Title: Neurofeedback for Tourette Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0206017435; R01MH095789 (NIH)
Record Dates: First submitted 2012-10-03; First posted 2012-10-05 (Estimated); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Tourette Syndrome; Chronic Tic Disorder
Keywords: neurofeedback; biofeedback; real-time fMRI; rt-fMRI; functional connectivity; fMRI
MeSH Terms: conditions — Tourette Syndrome; Tic Disorders | interventions — Neurofeedback; Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neurofeedback first (Experimental): Neurofeedback then sham feedback
  Interventions: Procedure: Neurofeedback; Procedure: Sham feedback
- Sham first (Experimental): Sham feedback then neurofeedback
  Interventions: Procedure: Neurofeedback; Procedure: Sham feedback

INTERVENTIONS:
Procedure: Neurofeedback
  Other Names: biofeedback; real-time fMRI biofeedback
Procedure: Sham feedback

SUMMARY:
The aim of this study is to train patients with tic disorders to control activity in a region of their brain that has been associated with the urge to tic. Patients will be given direct feedback regarding activity in this brain area while they are undergoing functional magnetic resonance imaging (fMRI) scanning, and will try to learn to control activity in the region during these feedback sessions. In separate sessions, patients will be given sham feedback based on the brain patterns of a prior subject rather than their own brain patterns. Our primary hypothesis is that the biofeedback training will reduce their tic symptoms more than the sham feedback.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tourette Syndrome or Chronic Tic Disorder
* currently active tics
* aged 11-19
* ability to execute most common tics without moving head while lying on back

Exclusion Criteria:

* Blindness (because feedback is provided visually)
* Lifetime diagnosis of pervasive developmental disorder, bipolar disorder, or psychotic disorder.
* Presence of any serious psychiatric or psychosocial condition requiring initiation of new treatment or change in current treatment.
* Neurological conditions affecting central nervous system, with the exception that predisposition to migraine will not be grounds for exclusion
* Change in medication in the month prior to beginning the study
* Unwillingness to keep medication stable over the course of the intervention
* Full braces (but some retainers are OK)
* Claustrophobia of a degree that they cannot comfortably be scanned
* If common tics involve dramatic changes in breathing that could alter blood oxygenation measurements
* Inability to keep head still while executing most common tics
* Inability to keep head still in mock scanner
* Inability or unwillingness to understand or follow the instructions
* Pregnancy or possible pregnancy
* Subjects may also be excluded after the first magnetic resonance scan if we are unable to localize a region of their supplementary motor area involved in tics - leaving us without a target area for biofeedback.

Ages: 11 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-10; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Tic severity | Tic severity assessed approximately half a week PRIOR TO beginning biofeedback/sham feedback.
  A modified version of the Yale Global Tic Severity Scale (YGTSS) will be used, that queries subjects regarding symptoms over the last 3 days (rather than the 2 week period used in the standard scale). Total YGTSS score on this modified scale will be used as the measure of tic severity.
Tic severity | Tic severity assessed approximately half a week AFTER completing biofeedback/sham feedback.
  A modified version of the Yale Global Tic Severity Scale (YGTSS) will be used, that queries subjects regarding symptoms over the last 3 days (rather than the 2 week period used in the standard scale). Total YGTSS score on this modified scale will be used as the measure of tic severity.

SECONDARY OUTCOMES:
Control over target brain area | Assessed approximately half a week BEFORE biofeedback/sham biofeedback.
  Control task scans will be conducted in which subjects are cued to alternately increase and decrease activity in their target area without receiving any feedback. The percent signal change in the BOLD signal in the target area during increase relative to decrease blocks will be used as the measure of control over the brain area.
Control over target brain area | Assessed approximately half a week AFTER biofeedback/sham biofeedback.
  Control task scans will be conducted in which subjects are cued to alternately increase and decrease activity in their target area without receiving any feedback. The percent signal change in the BOLD signal in the target area during increase relative to decrease blocks will be used as the measure of control over the brain area.

OTHER OUTCOMES:
Functional connectivity patterns in the brain | Assessed approximately half a week BEFORE biofeedback/sham biofeedback.
  Functional connectivity will be assessed based on temporal correlations in resting state functional imaging data.
Functional connectivity patterns in the brain | Assessed approximately half a week AFTER biofeedback/sham biofeedback.
  Functional connectivity will be assessed based on temporal correlations in resting state functional imaging data.
Clinical improvement | Clinical improvement will be assessed approximately half a week AFTER biofeedback/sham feedback
  The Clinical Global Impression - Improvement scale will be used to assess improvement over the course of the biofeedback/sham feedback

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hampson, Ph.D., Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States